CLINICAL TRIAL: NCT07203807
Title: Methodological Study on the Minimum Number of Blocks in fNIRS: Brain Activity During Voluntary Movement and During Illusory Movement Induced by Vibratory Tendon Stimulation of the Right Distal Upper Limb in Healthy Right-handed Participants
Brief Title: Study of the Optimal Number of Repetitions to Investigate the Cerebral Activity by fNIRS During a Voluntary Movement and an Illusory Movement Induced by Vibration
Acronym: MoViBloc
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Régional d'Orléans (Other)
Responsible Party: Sponsor
Other Study IDs: CHUO-2025-17
Record Dates: First submitted 2025-09-25; First posted 2025-10-02 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Healthy
Keywords: fNIRS; Blocks; Movement; Illusion
MeSH Terms: conditions — Bites and Stings; Illusions

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy young: Healthy young participants aged 18 to 40
  Interventions: Other: Voluntary movement and illusory movement of the right upper limb induced by TVS.

INTERVENTIONS:
Other: Voluntary movement and illusory movement of the right upper limb induced by TVS. — The protocol comprises two different modalities: Voluntary movement and illusory movement of the right upper limb induced by TVS.
  The experiment will begin and end with a one-minute rest period. Participants will be asked to open and close their right hand 20 times in 10 seconds. Similarly, they will experience 10 seconds of TVS-induced illusory movement 20 times. Each task epoch will be preceded by a 12-20 second resting period.
  Both conditions will be randomized and counterbalanced. Participants can start with either the voluntary movement task or the illusory.

SUMMARY:
The purpose of this study is to investigate the cerebral activation of healthy participants during a voluntary movement and an illusory movement induced by vibration.

This will be done by repeating both tasks 20 times for 10 seconds.

The study aims to determine the minimum number of repetitions (blocks) required to maximize cerebral activity.

DETAILED DESCRIPTION:
Functional near-infrared spectroscopy (fNIRS) is a non-invasive method that measures cortical hemodynamic responses by measuring variations in oxyhemoglobin (HbO) and deoxyhemoglobin (HbR). Thanks to its portability, ease of use, and low cost, fNIRS is particularly well suited to the study of neurological populations such as stroke patients.

To obtain a robust hemodynamic response, fNIRS studies use a block-design experimental paradigm, alternating between periods of task performance and rest. However, there is considerable heterogeneity in the number of blocks used in the literature, making it difficult to construct an optimal paradigm. Among the methodological issues, knowledge of the minimum number of blocks for which the cerebral response is maximal appears to be a key point.

It is generally acknowledged that increasing the number of blocks reduces intra-individual variability and improves the detection of task-specific responses. However, increasing the number of blocks increases the acquisition time, which can lead to fatigue or discomfort, particularly in elderly participants or participants with neurological disorders. A compromise must be found between methodological precision and clinical tolerance in the construction of future experimental paradigms, particularly those involving a motor task in a neurological rehabilitation context.

To date, the literature does not recommend a specific number of blocks based on the actual motor task (voluntary movement) or illusory task (induced by tendon vibration stimulation (TVS)), as both modalities are used in rehabilitation. Improving our understanding of the relationship between the number of blocks and the hemodynamic response measured by fNIRS depending on the type of task would enable us to move towards standardizing experimental paradigms.

The aim of this study is to identify the minimum number of blocks required to obtain a maximal cerebral hemodynamic response (variations in HbO and HbR), measured by fNIRS during a unilateral hand motor task and an illusory movement induced by TVS in healthy participants. Ultimately, these results will help optimize fNIRS experimental paradigms by ensuring reliable capture of task-related brain activity in a minimum of time, compatible with a pathological population.

The protocol comprises two different modalities: Voluntary movement and illusory movement of the right upper limb induced by TVS. This experiment will be conducted on young, healthy participants aged 18 to 40.

The experiment will begin and end with a one-minute rest period. Participants will be asked to open and close their right hand 20 times in 10 seconds. Similarly, they will experience 10 seconds of TVS-induced illusory movement 20 times. Each task epoch will be preceded by a 12-20 second resting period.

Both conditions will be randomized and counterbalanced. Participants can start with either the voluntary movement task or the illusory.

The fNIRS devices that will be used are the Brite MKII and Brite MKIII (Artinis Medical Systems, the Netherlands).

The vibration tool is a VibraMoov vibrator from Technoconcept in Mane, France.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy volunteers aged 18 to 40
2. Right-handed: Edinburgh laterality test short format QL > 60 (Veale et al., 2014).
3. Sufficient command of the French language to understand instructions
4. No known neurological medical history

Exclusion Criteria:

1. Allergy to neoprene (fNIRS cap material)
2. Hair volume preventing the cap from fitting and/or access to the scalp
3. Injury to right upper limb causing pain during mobilization
4. Protected person (under guardianship or trusteeship)
5. Person under court protection
6. Persons deprived of liberty
7. Persons not affiliated to a social security scheme
8. Pregnant or breast-feeding women
9. Volunteers opposed to the study

Ages: 18 Years to 40 Years | Sex: All
Age Groups: Adult
Study Population: Healthy young adult aged 18 to 40
Sampling Method: Non-Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2025-10-27 (Actual); Primary Completion 2025-10-31 (Actual); Study Completion 2025-10-31 (Actual)

PRIMARY OUTCOMES:
Cerebral hemodynamic variations in the sensorimotor areas assessed by fNIRS with 42 long channels and 4 short channels. | Day 0
  HbO will be considered as the primary outcome measure of the cerebral activity through the hemodynamic response
Cerebral hemodynamic variations in the frontoparietal areas assessed by fNIRS with 42 long channels and 4 short channels | Day 0
  HbO will be considered as the primary outcome measure of the cerebral activity through the hemodynamic response

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Orléans, Orléans, France

REFERENCES:
- [Background] Edin BB, Vallbo AB. Dynamic response of human muscle spindle afferents to stretch. J Neurophysiol. 1990 Jun;63(6):1297-306. doi: 10.1152/jn.1990.63.6.1297. PMID 2141632
- [Background] Herold F, Wiegel P, Scholkmann F, Thiers A, Hamacher D, Schega L. Functional near-infrared spectroscopy in movement science: a systematic review on cortical activity in postural and walking tasks. Neurophotonics. 2017 Oct;4(4):041403. doi: 10.1117/1.NPh.4.4.041403. Epub 2017 Aug 1. PMID 28924563
- [Background] Naito E, Morita T, Amemiya K. Body representations in the human brain revealed by kinesthetic illusions and their essential contributions to motor control and corporeal awareness. Neurosci Res. 2016 Mar;104:16-30. doi: 10.1016/j.neures.2015.10.013. Epub 2015 Nov 10. PMID 26562333
- [Background] Pinti P, Tachtsidis I, Hamilton A, Hirsch J, Aichelburg C, Gilbert S, Burgess PW. The present and future use of functional near-infrared spectroscopy (fNIRS) for cognitive neuroscience. Ann N Y Acad Sci. 2020 Mar;1464(1):5-29. doi: 10.1111/nyas.13948. Epub 2018 Aug 7. PMID 30085354
- [Background] Schneider C, Marquis R, Johr J, Lopes da Silva M, Ryvlin P, Serino A, De Lucia M, Diserens K. Disentangling the percepts of illusory movement and sensory stimulation during tendon vibration in the EEG. Neuroimage. 2021 Nov 1;241:118431. doi: 10.1016/j.neuroimage.2021.118431. Epub 2021 Jul 28. PMID 34329723